CLINICAL TRIAL: NCT04823442
Title: Sympathomimetics and Sympatholytics in Type 2 Diabetes: Teaching Old Drugs New Tricks
Brief Title: Activation of Brown Adipose Tissue Metabolism Using Mirabegron
Acronym: GB9
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Laval University (Other)
Responsible Party: Principal Investigator, Denis Blondin, Assisant professor, Université de Sherbrooke
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2021-3791
Record Dates: First submitted 2021-03-26; First posted 2021-03-30 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — mirabegron; Bisoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study A (Active Comparator): Metabolic PET study with mirabegron
  Interventions: Drug: Mirabegron
- Study B (Experimental): Metabolic PET study with mirabegron and bisoprolol
  Interventions: Drug: Mirabegron; Drug: Bisoprolol Fumarate

INTERVENTIONS:
Drug: Mirabegron — Mirabegron: a single dose of 200 mg mirabegron (4 tablets of 50 mg)
  Other Names: Myrbetriq
Drug: Bisoprolol Fumarate — a single dose of 10 mg (2 tablets of 5 mg)
  Other Names: Apo Bisoprolol
  Arms: Study B

SUMMARY:
Could sympathomimetics and sympatholytics drugs safe for the management of Type 2 Diabetes (T2D)? Based on recent evidence, we propose that pharmacological stimulation of Beta-3 adrenergic receptor (ADBR3) at higher doses of Mirabegron may be required to elicit changes in glycemia, but should be combined with Beta-1 adrenergic receptor (ADRB1) antagonists to suppress the unwanted effects on the cardiovascular system.

Together, several results establish a previously unappreciated cross-talk between Gs-coupled ADRB1 and ADRB3 in adipose tissue for the control of glucose homeostasis. Moreover, these data suggest that antagonizing ADRB1 may be a good way to significantly lower the dose of ADRB3 agonist required for glucose control.

Therefore, we believe that there are therapeutic opportunities in targeting adrenergic receptors for the treatment of T2D at least in young/middle aged people.

DETAILED DESCRIPTION:
In brief, participants will take part in 2 metabolic studies (A and B) performed in random order and at an interval of 7 to 14 days. Each metabolic study will last 8.5 hours with a baseline period of 2.5 hours. Participants will ingest either 200 mg of the ADRB3 agonist mirabegron (Myrbetriq, Astellas Pharma Canada) alone (study A) or in combination with 10 mg of bisoprolol, an ADRB1-antagonist (study B), at time 0.

The radioactive PET tracers (PET: positron emission tomography) used in this study are the [11C]-acetate and [18F]-FDG to estimate BAT oxidative metabolism and glucose metabolism, respectively. The perfusion of [6,6 D2]-glucose, [1,1,2,3,3-2H]-glycerol and [U-13C]-palmitate stable isotopes will also be performed in this study from time -150 min. to +300 min to examine the systemic appearance rate of glucose, glycerol and fatty acids, respectively. These studies will be almost identical (same perfusion of stable and radioactive tracers, same number of PET acquisitions) except for the drug which will be administered orally at time 0.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with normal glucose tolerance determined according to an oral glucose tolerance test;
* BMI ≤ 30 kg/m2.

Exclusion Criteria:

* Plasma triglycerides > 5.0 mmol/L at fasting;
* More than 2 alcohol consumption per day;
* More than 1 cigarette per day;
* History of total cholesterol level > 7 mmol/L, of cardiovascular disease, hypertensive crisis;
* Treatment with fibrates, thiazolidinedione, insulin,betablockers or other drugs with effects on insulin resistance or lipid metabolism (exception for antihypertensive drugs, statins or metformin);
* Presence of a noncontrolled thyroid disease, renal or hepatic disease, history of pancreatitis, bleeding diatheses, cardiovascular disease or any other serious medical conditions;
* History of serious gastrointestinal disorders (malabsorption, peptic ulcer, gastroesophageal reflux having required a surgery, etc.); reflux having required a surgery, etc.);
* Presence of a pacemaker;
* Have undergone of PET study or CT scan in the past year;
* Chronic administration of any medication;

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
Change in activation of Brown Adipose Tissue (BAT) (oxidative metabolism and blood flow) | 30 minutes before and 210 minutes after drug administration
  Measured with 11C-acetate using dynamic PET/CT acquisition.
BAT glucose uptake | 240 minutes after drug administration
  Assessed using i.v. injection of 18FDG with sequential dynamic PET/CT scanning

SECONDARY OUTCOMES:
Whole-body glucose partitioning | 300 minutes after drug administration
  Assessed using i.v. injection of 18FDG with static PET/CT scanning
Whole-body lipolysis | 150 minutes before and mean of time 180, 240 and 300 minutes after drug administration (steady state).
  Systemic appearance rate of glycerol and fatty acid determined by perfusion of [1,1,2,3,3-2H]-glycerol, [U-13C]-palmitate tracers. and concentration of total NEFA, triglycerides, palmitate, oleate, linoleate, glycerol.
Hepatic Glucose production | 150 minutes before and mean of time 180, 240 and 300 minutes after drug administration (steady state).
  Systemic appearance rate of glucose determined by perfusion of [6,6 D2]-glucose
Substrate utilisation | 150 minutes before and mean of time 210 and 270 minutes after drug administration (steady state).
  VO2 and VCO2 will be measured by indirect calorimetry to calculate carbohydrate and fatty acid oxidation rates.
BAT lipolysis | baseline and 300 minutes after drug administration
  Estimated by quantifying changes in tissue radiodensity with CT.
Changes in pancreatic and gut hormones | 150 minutes before and mean of time 180, 240 and 300 minutes after drug administration (steady state).
  measured with ELISA and Milliplex.

CONTACTS AND LOCATIONS:
Overall Officials: Denis Blondin, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de recherche du CHUS, Sherbrooke, Quebec, Canada

REFERENCES:
- [Result] Dumont L, Caron A, Richard G, Croteau E, Fortin M, Frisch F, Phoenix S, Dubreuil S, Guerin B, Turcotte EE, Carpentier AC, Blondin DP. The effects of the beta1-adrenergic receptor antagonist bisoprolol administration on mirabegron-stimulated human brown adipose tissue thermogenesis. Acta Physiol (Oxf). 2024 May;240(5):e14127. doi: 10.1111/apha.14127. Epub 2024 Mar 19. PMID 38502056
- [Derived] Chunchai T, Chinchapo T, Sripetchwandee J, Thonusin C, Chattipakorn N, Chattipakorn SC. Lipopolysaccharide exacerbates depressive-like behaviors in obese rats through complement C1q-mediated synaptic elimination by microglia. Acta Physiol (Oxf). 2024 May;240(5):e14130. doi: 10.1111/apha.14130. Epub 2024 Mar 10. PMID 38462756
- See also: publication of results — https://pubmed.ncbi.nlm.nih.gov/38502056/